CLINICAL TRIAL: NCT00049907
Title: Cardiac and Renal Disease Study (CARDS)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1200; R01HL071074 (NIH)
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2006-01

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Cerebrovascular Accident; Heart Failure; Heart Diseases; Peripheral Vascular Diseases; Diabetes Mellitus; Hypertension; Kidney Failure, Chronic
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Stroke; Heart Failure; Heart Diseases; Peripheral Vascular Diseases; Diabetes Mellitus; Hypertension; Kidney Failure, Chronic

SUMMARY:
To examine the epidemiology of renal disease and its relationship to cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Mild-to-moderate chronic renal insufficiency (CRI) has been reaching epidemic proportions in the United States. Studies relating mild-to-moderate chronic renal insufficiency and cardiovascular risk were limited and inconsistent. Although much had been learned about the natural history and adverse outcomes associated with end-stage renal disease (ESRD), there was little specific information regarding risk factors for the development or progression of renal disease.

The study was initiated in response to a Request for Applications entitled "NHLBI Innovative Research Grant Program" released in July, 2001. The purpose of the initiative was to support new approaches to heart, lung, and blood diseases and sleep disorders that used existing data sets or existing biological specimen collections whether obtained through National Heart, Lung, and Blood Institute support or not.

DESIGN NARRATIVE:

The population-based study used data on an ethnically diverse large cohort of male and female health plan enrollees with extended follow-up. The study evaluated: a) whether baseline and decline in renal function over time were independent predictors of coronary heart disease (CHD), stroke, heart failure and peripheral vascular disease; b) effect modifiers of these relationships,including baseline hypertension and diabetes status. The study determined whether baseline and increase over time in blood pressure level (as well as prevalent and incident hypertension) were predictive of the subsequent risk of ESRD after adjusting for diabetes and for baseline serum creatinine, proteinuria and hematuria. The study also examined other potential predictors of ESRD including demographic factors (race/ethnicity, level of education) total cholesterol level, family history of renal disease, body mass index, sagittal abdominal diameter, cigarette (as well as cigar and pipe) smoking, coffee intake, alcohol consumption, family history of renal disease and self-reported occupational exposures. The study used existing longitudinal data resources at the Northern California Kaiser Permanente Division of Research and available patient-level cross-linkage with the US Renal Data System end-stage renal disease registry to obtain comprehensive renal and cardiovascular outcomes.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Iribarren — Kaiser Foundation Research Institute

REFERENCES:
- [Background] Hsu CY, McCulloch CE, Darbinian J, Go AS, Iribarren C. Elevated blood pressure and risk of end-stage renal disease in subjects without baseline kidney disease. Arch Intern Med. 2005 Apr 25;165(8):923-8. doi: 10.1001/archinte.165.8.923. PMID 15851645
- [Background] Hsu CY, McCulloch CE, Iribarren C, Darbinian J, Go AS. Body mass index and risk for end-stage renal disease. Ann Intern Med. 2006 Jan 3;144(1):21-8. doi: 10.7326/0003-4819-144-1-200601030-00006. PMID 16389251